CLINICAL TRIAL: NCT06551558
Title: Impact of a Global Warming Strategy, From the Patient Arrival in the Operating Room to His Discharge From the Recovering Room, Versus a Recommended Management of Intraoperative Warming on the Prevalence of Hypothermia in the Recovering Room
Brief Title: Impact of a Global Warming Strategy of the Patient on the Prevalence of Hypothermia in the Recovering Room
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RéGlo
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-06

CONDITIONS: Hypothermia; Anesthesia; Perioperative/Postoperative Complications
MeSH Terms: conditions — Hypothermia; Postoperative Complications | interventions — Global Warming

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RéGlo arm (Experimental): Innovative support with global warming strategy.
  Interventions: Other: global warming
- Control arm (Other): Support according to recommendations
  Interventions: Other: per operative warming

INTERVENTIONS:
Other: global warming — A systematic pre- and post-operative warming associated with the optimization of per-operative warming.
  Arms: RéGlo arm
Other: per operative warming — per-operative warming only thanks to the "Optimized" Forced air blanket with a prewarming of 10 minutes performed in the operating room.
  Arms: Control arm

SUMMARY:
50% of patients are hypothermic when they arrive in the recovery room. This hypothermia is potentially at risk for the patient (increases bleeding, risk of infection, risk of cardiac involvement, morbid mortality) and 33,2% steel hypothermic when they discharge from the recovering room. The anesthesia team must prevent these risks through prevention and treatment measures. Currently the majority of patient warming is done only in the operating room, we want to measure the impact of the extension of this warming before and after the surgery on the patient's temperature and on side effects related to hypothermia.

DETAILED DESCRIPTION:
Hypothermia is defined as a core temperature below 36°C. It is classified by severity stage. A temperature below 36°C is mild hypothermia, below 35°C moderate hypothermia and below 34°C severe hypothermia.

The impact of hypothermia on the body is related to decreased metabolic and immune activities. The vasoconstriction induced by hypothermia implies a decrease in vascularization of the organs that can cause tissue damage.

These effects explain the role of hypothermia in the pathophysiology of certain perioperative and postoperative complications in the longer term.

Intraoperative hypothermia is responsible for the increase of:

* 4 times the risk of Surgical Site Infection,
* twice the risk of cardiovascular morbidity, associated with increased mortality,
* 33% of transfusion need,
* 1.5 times the need for continued mechanical ventilation,
* 3 times the duration of recovering room,
* twice the hospital stay. This is why hypothermia is responsible for excess perioperative mortality.

According to a 2019 study (Alfonsi P, Bekka S, Aegerter P, SFAR Research Network investigators. Prevalence of hypothermia on admission to recovery room remains high despite a large use of forced-air warming devices: Findings of a non-randomized observational multicenter and pragmatic study on perioperative hypothermia prevalence in France), the prevalence of hypothermia increases from 16.2% of patients before anesthetic induction to 53.5% of patients admitted to the Recovering room. At the end of Recovering room, 33.2% of patients were hypothermic. Among these patients, 15.2% became hypothermic during the recovering room stay.

The risk factors for perioperative hypothermia are multiple:

Patient-related factors: low body mass index; undernutrition; ASA score > 1; pre-existing conditions altering thermoregulation (ex: diabetes with polyneuropathy, hypothyroidism, consumption of sedative or psychoactive drugs); pre-existing hypothermia at surgery.

Factors related to anesthesia techniques: duration of anesthesia > 2 hours; combined general and neuro-axial anesthesia; administration of large volumes of intravenous solutes or transfusion of non-rewarmed globular units.

Factors related to surgery: type, extent and duration of surgery witch use of large amounts of unheated irrigation fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing laparoscopic visceral surgery under general anesthesia with transition to recovering room

Exclusion Criteria:

* Patient undergoing urgent surgery.
* Presence of pre-existing infection (temperature higher than 38°C when receiving the patient in the hospital ward.
* Patient with predetermined length of stay in recovering room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, the prevalence of hypothermia at the exit of Interventional for patients who underwent laparoscopic visceral surgery. | 1 day
  Proportion of patients with hypothermia after discharge of recovering room. Hypothermia is defined as a body temperature < 36°C.

SECONDARY OUTCOMES:
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, the average total mechanical ventilation time | 1 day
  it is the time between intubation and extubation, expressed in minutes.
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, the average thermal comfort of preoperative patients, on arrival in the pre- anesthesia room | 1 day
  evaluated by the Likert scale, ranging from 0 for discomfort too cold with strong chills to 4 for discomfort too hot with sweat with optimal comfort to 2 (self-assessment)
Compare between the experimental group of global warming (RéGlo) and the control group of per- operative warming, the average thermal comfort of preoperative patients, on arrival in the recovering room | 1 day
  every 15minutes until discharge, evaluated by the Likert scale, ranging from 0 for discomfort too cold with strong chills to 4 for discomfort too hot with sweat with optimal comfort to 2 (self-assessment).
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, the proportion of patients in intraoperative hypothermia | 1 day
  number of patient with body temperature under 36°C between arrival in pre-operative room and discharge of operating room
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, The average time spent below 36°C (mild hypothermia) | 1 day
  expressed in minutes.
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, The average time spent below 35°C (moderate hypothermia) | 1 day
  expressed in minutes.
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, The average time spent below 34°C (severe hypothermia) | 1 day
  expressed in minutes.
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, The lowest average temperature reached in °C over the entire management | 1 day
  the lowest temperture between arrival in the pre-anaesthesia room and exit from recovering room
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, The proportion of hypothermic patients arriving in recovering room | 1 day
  number of patient with a temperature below 36°C
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, The average duration of oxygen therapy | 1 day
  calculated from the introduction of oxygen therapy until its withdrawal in post extubation, regardless of the time of implementation or cessation before resumption of treatment (failure to withdraw oxygen therapy will not be considered), expressed in minutes.
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, Post-intervention complications in recovering room, the average number of Nausea or Vomiting Postoperative | 1 day
  number of patient with Nausea or Vomiting in recovering room evaluated every 15 minutes until discharge
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, Post-intervention complications in recovering room, the average number of chills | 1 day
  number of chills during post-operative monitoring by a Likert scale
Compare between the experimental group of global warming (RéGlo) and the control group of per-operative warming, Post-intervention complications in recovering room, the average number of stirring phase presence | 1 day
  number of stirring phase evaluated every 15 minutes until discharge
The average amount of blood loss per operation | 1 day
  blood loss measured from the time of entry into the operating theatre to the exit from the operating theatre expressed in millilitres.
The average of immediate post-operative blood loss | 1 day
  blood loss measured in recovering room expressed in millilitres
The general average of the thermal variation | 1 day
  the difference between the patient's lowest and highest temperature between their arrival in the pre-anaesthesia room and their exit from recovering room, expressed in degrees Celsius
The average of thermal variation in pre operative | 1 day
  the difference between the lowest and highest temperature of the patient between the arrival in the waiting room of the operating room and the arrival in the operating room, expressed in degrees Celsius
The average thermal variation in per operative | 1 day
  the difference between the lowest and highest temperature of the patient between the arrival and exit of the operating room, expressed in degrees Celsius
the average thermal variation in post operative | 1 day
  the difference between the lowest and highest temperature of the patient between arrival in and validation exit criteria of recovering room,expressed in degrees Celsius
The average length of stay in recovering room | 1 day
  difference between the time of arrival in recovering room and the time of obtaining the exit criteria , expressed in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Boisson, Pu-Ph, Principal Investigator — Poitiers University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfonsi P, Bekka S, Aegerter P; SFAR Research Network investigators. Prevalence of hypothermia on admission to recovery room remains high despite a large use of forced-air warming devices: Findings of a non-randomized observational multicenter and pragmatic study on perioperative hypothermia prevalence in France. PLoS One. 2019 Dec 23;14(12):e0226038. doi: 10.1371/journal.pone.0226038. eCollection 2019. PMID 31869333